CLINICAL TRIAL: NCT00282997
Title: A 12-Week, Open-Label, Safety Trial Of Pregabalin In Patients With Fibromyalgia
Brief Title: A Safety Study Of Pregabalin In Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081078
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2007-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin

SUMMARY:
To evaluate the safety of pregabalin in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the ACR criteria for fibromyalgia (ie, widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites.
* Patients must complete the double-blind study.

Exclusion Criteria:

* Patients who experienced a serious adverse event during the previous fibromyalgia study, which was determined to be related to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2006-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of pregabalin in patients with fibromyalgia

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- United States (72):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Pismo Beach, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Kenner, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Goose Creek, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Summerville, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Georgetown, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Killeen, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Woodstock, Vermont
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Arnold LM, Emir B, Murphy TK, Zeiher BG, Pauer L, Scott G, Petersel D. Safety profile and tolerability of up to 1 year of pregabalin treatment in 3 open-label extension studies in patients with fibromyalgia. Clin Ther. 2012 May;34(5):1092-102. doi: 10.1016/j.clinthera.2012.03.003. Epub 2012 Apr 14. PMID 22503162
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081078&StudyName=A+Safety+Study+Of+Pregabalin+In+Fibromyalgia